CLINICAL TRIAL: NCT05044884
Title: Effects of Otago Exercise Program vs Circuit Training on Balance in Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Effects of Otago Exercise Program vs Circuit Training on Balance in Chronic Obstructive Pulmonary Disease Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00960 Saba Nadeem
Record Dates: First submitted 2021-09-01; First posted 2021-09-16 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: COPD
Keywords: Chronic obstructive pulmonary disease (COPD); Pulmonary rehabilitation; Balance; Otago exercise; Circuit training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago exercise group (Experimental): The Otago exercise group will practice the Otago exercise protocol which includes strength and balance exercises along with pulmonary rehabilitation.
  * 3 times per week for 8 weeks.
  * Each session will be of 60 minutes
  * Total number of sessions: 24
  Interventions: Other: Otago Exercise training
- Circuit training group (Active Comparator): The Circuit training group will practice balance exercises including Stance exercise, Functional strength exercise, Transition exercise and Gait training along with pulmonary rehabilitation.
  * 3 times per week for 8 weeks.
  * Each session will be of 60 minutes
  * Total number of sessions: 24
  Interventions: Other: Circuit training

INTERVENTIONS:
Other: Otago Exercise training — 1. Warm-up exercises. Chair March, Arm swings ( 30 second), Head movement, neck movement, back extension, trunk movement, ankle movement (repeat 5 times).
     Back of thigh stretch, calf stretch, (hold for 8 seconds).
  2. Strengthening exercises Front knee strengthening, back knee strengthening, side hip strengthening (2 or more sets of 10 reps) Calf raises, toe raises (repeat this exercises 10 to 20 times)
  3. Balance improvement exercises Knee bends, heel-toe standing, heel toes walking, one leg stand ( start with 5 sec move up to 10 sec) Side walk, heel walking, sit to stand, backwards walking, heel toes walking backwards, walking and turning around, stair walking (10 steps).
  4. Cool-down session Back of thigh stretch, calf stretches ( 10 to 20 sec hold, 1 to 3 reps)
  5. Pulmonary rehabilitation program
     * Daily breathing exercises (e.g. diaphragmatic, pursed lip breathing).
     * Stretch exercise for major respiratory muscles.
  Arms: Otago exercise group
Other: Circuit training — 1. Functional strength exercises Heel raise, toe raise, walking on toes, step ups in all directions ( forward, backward and sideways) (2 sets and 8 reps)
  2. Stance exercises Tandem, narrow, one leg stance, and stand on uneven surfaces with open eyes (each exercise 30 seconds) Tandem, narrow, one leg stance, and stand on uneven surfaces with eyes closed (each exercise 15seconds).
  3. Transition exercises Sit to stand from chair with arms (10 reps) and then without arms support (5 reps).
     Sit on floor and stand up with assistance and then without assistance.
  4. Gait training Walking tandem, sideway and backward with arm support. Walking tandem, sideway and backward without arm support Walking tandem, sideway and backward over obstacles
  5. Pulmonary rehabilitation program
     * Daily breathing exercises (e.g. diaphragmatic, pursed lip breathing).
     * Stretch exercise for major respiratory muscles
  Arms: Circuit training group

SUMMARY:
The study is designed to compare circuit training and otago exercise program for improvement of balance in COPD patients. Although both techniques are effective for balance training but Otago exercise program is home-based exercise program, which, if proven effective, will help the COPD patients to do work up at home, thereby reducing cost of hospital visits and improving balance ability and thus the quality of life more effectively.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a respiratory disease that result in progressive restriction of airflow and respiratory distress and is the 4th leading cause of death. In specific, it happens among smokers over the age of 40 and individuals exposed to biomass smoke. The prevalence of COPD is expected to increase as the population ages. Pakistan is a lower-middle-income country, and facing a high burden of chronic obstructive pulmonary diseases. The prevalence of COPD among Pakistani adults aged more than 40 years is 2.1% In addition to pulmonary symptoms, patients with chronic obstructive pulmonary disease develop many other manifestations of the disease, such as cardiovascular co morbidities, peripheral muscle dysfunction, weight loss, systemic inflammation, and psychological problems. People also have reduced capacity for exercise and functional mobility. Among all, one important extra respiratory manifestation is impaired balance. It is a frequent problem in stable COPD and increases with the severity of the disease. As in COPD there is loss of body cells which causes skeletal muscle weakness and balance impairment.

Since skeletal muscle dysfunction in people with COPD is a commonly identified impairment, it is not surprising that lower-limb muscle weakness has also been linked in this population to balance deficits and increased risk of falling. Muscle strength in both the upper and lower extremities is reduced in COPD patients along with impairments in exercise tolerance.

Pulmonary rehabilitation (PR) is an effective COPD intervention that involves exercise training and psychosocial support, and patient education to achieve maximum community independence and function. This recommended standard of care, however, focuses primarily on training peripheral muscles through endurance and strength training and does not include a particular training component. The effective intervention to successfully reduce both the rate and risk of falling has been shown to be exercise with balance-specific training.

As COPD decreases the amount of physical activity, even early in the disease phase, and impairs the strength of the lower limb muscle thus affecting balance. Balance training protocols together with pulmonary rehabilitation exercises helps to improve balance and symptoms of COPD. Although both circuit training and Otago exercise program are effective for balance training but Otago exercise program is home-based exercise program, which, if proven effective, will help the COPD patients to do work up at home, thereby reducing cost of hospital visits and improving balance ability and thus the quality of life more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients.
* Patients with mild / moderate COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.
* Patients with fall history in the past 5 years.

Exclusion Criteria:

* Oxygen-dependent or mechanically ventilated patients.
* Patients with impaired hearing or cognition, (e.g., dementia or neurological condition)
* Patients with limited balance and mobility owing musculoskeletal or neurological condition.
* Patients with unstable cardiovascular disease.
* Patients with intellectual disabilities.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 8 weeks
  Berg Balance Scale was originally developed to measure balance in the elderly, it has since been used to measure balance in a wide variety of patients. Each of these items is scored from 0 to 4, which are summed to make a total score between 0 and 56, with a higher score indicating better balance. The relative intrarater reliability of the Berg Balance Scale is 0.98 (0.97 to 0.99). Relative inter-rater reliability is 0.97 (0.96 to 0.98). Changes in berg balance scale from baseline to 4th and after 8 weeks of intervention will be assessed.
Unipedal Stance (UPST) test | 8 weeks
  The Unipedal stance test is described as a method of quantifying static balance ability and is useful in explaining other variables of importance such as frailty and self-sufficiency in activities of daily living, gait performance, and fall status. It can be used in a variety of settings and requires minimal equipment or training. It is a valid measure. Abnormal unipedal stance test (UPST) time with the eyes open is related to conditions such as peripheral neuropathy and intermittent claudication. Decreased eyes open UPST time is also associated with an increased risk for falls. Its inter-rater reliability was determined to be excellent with an intra-class correlation coefficient of 0.994(95% confidence interval 0.989-0.996) for eye open and 0.998 (95% confidence interval 0.996-0.999) for eye close. Average time of unipedal stance in healthy older adults is < 10 seconds. Changes in UPST from baseline to 4th and after 8 weeks of intervention will be assessed.

SECONDARY OUTCOMES:
St. George Respiratory questionnaire for quality of life (QOL) | 8 weeks
  The most commonly used disease-specific quality of life measure for COPD patients is the St. George's Respiratory Questionnaire (SGRQ). Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.. It is divided in two parts. Part I produces the Symptoms score, and Part 2 the Activity and Impacts scores. The reliability coefficient was 0.94 for the overall scale and 0.72 for "Symptoms", 0.89 for "Activity", and 0.89 for "Impacts" subscales.
  A total score is calculated from 0 (no health impairment) to 100 (maximum health impairment) Changes in St. George Respiratory questionnaire for quality of life from baseline to 4th and after 8 weeks of intervention will be assessed.
Peak expiratory flow rate (PEFR) | 8 weeks
  Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings. Changes in PEFR from baseline to 4th and after 8 weeks of intervention will be assessed.
Forced vital capacity (FVC) | 8 weeks
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal. Changes in FVC from baseline to 4th and after 8 weeks of intervention will be assessed.
Forced expiratory volume in 1sec (FEV1) | 8 weeks
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal. Changes in FEV1 from baseline to 4th and after 8 weeks of intervention will be assessed.
FVC/FEV1 | 8 weeks
  FVC/FEV1 measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65). Changes in FEV1/FVC from baseline to 4th and after 8 weeks of intervention will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Suman Sheraz, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crisan AF, Oancea C, Timar B, Fira-Mladinescu O, Tudorache V. Balance impairment in patients with COPD. PLoS One. 2015 Mar 13;10(3):e0120573. doi: 10.1371/journal.pone.0120573. eCollection 2015. PMID 25768731
- [Background] Beauchamp MK, Brooks D, Ellerton C, Lee A, Alison J, Camp PG, Dechman G, Haines K, Harrison SL, Holland AE, Marques A, Moineddin R, Skinner EH, Spencer L, Stickland MK, Xie F, Goldstein RS. Pulmonary Rehabilitation With Balance Training for Fall Reduction in Chronic Obstructive Pulmonary Disease: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Nov 20;6(11):e228. doi: 10.2196/resprot.8178. PMID 29158206
- [Background] de Castro LA, Ribeiro LR, Mesquita R, de Carvalho DR, Felcar JM, Merli MF, Fernandes KB, da Silva RA, Teixeira DC, Spruit MA, Pitta F, Probst VS. Static and Functional Balance in Individuals With COPD: Comparison With Healthy Controls and Differences According to Sex and Disease Severity. Respir Care. 2016 Nov;61(11):1488-1496. doi: 10.4187/respcare.04749. Epub 2016 Aug 2. PMID 27484106
- [Background] Porto EF, Castro AA, Schmidt VG, Rabelo HM, Kumpel C, Nascimento OA, Jardim JR. Postural control in chronic obstructive pulmonary disease: a systematic review. Int J Chron Obstruct Pulmon Dis. 2015 Jun 29;10:1233-9. doi: 10.2147/COPD.S63955. eCollection 2015. PMID 26170652
- [Background] Marques A, Jacome C, Cruz J, Gabriel R, Figueiredo D. Effects of a pulmonary rehabilitation program with balance training on patients with COPD. J Cardiopulm Rehabil Prev. 2015 Mar-Apr;35(2):154-8. doi: 10.1097/HCR.0000000000000097. PMID 25517104
- [Background] Dadgari A, Aizan Hamid T, Hakim MN, Chaman R, Mousavi SA, Poh Hin L, Dadvar L. Randomized Control Trials on Otago Exercise Program (OEP) to Reduce Falls Among Elderly Community Dwellers in Shahroud, Iran. Iran Red Crescent Med J. 2016 Feb 14;18(5):e26340. doi: 10.5812/ircmj.26340. eCollection 2016 May. PMID 27478629